CLINICAL TRIAL: NCT06523595
Title: A Phase 1, Open-label Study Evaluating the Pharmacokinetic Drug-drug Interactions Between VX-993 and Metformin in Healthy Adult Subjects
Brief Title: Evaluation of the Pharmacokinetic Drug-drug Interactions Between VX-993 and Metformin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX24-993-006
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-993 and Metformin (Experimental): Metformin will be administered to participants as a single oral dose on Day 1 and then co-administered with VX-993 on Day 10. VX-993 dose will be administered every 12 hours (q12h) from Day 5 through Day 14.
  Interventions: Drug: VX-993; Drug: Metformin

INTERVENTIONS:
Drug: VX-993 — Suspension for Oral Administration.
Drug: Metformin — Tablets for Oral Administration.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic drug-drug interactions, safety, and tolerability of co-administration of VX-993 and metformin in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 Kilogram per square meter (kg/m^2)
* A total body weight of more than (>) 50 Kg
* Nonsmoker or ex-smoker for at least 3 months before the first study drug dose

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Metformin in Absence and Presence of VX-993 | From Day 1 up to Day 14
Area Under the Concentration Versus Time Curve for the Last Measurable Concentration (AUClast) of Metformin in Absence and Presence of VX-993 | From Day 1 up to Day 14
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of Metformin in Absence and Presence of VX-993 | From Day 1 up to Day 14

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 29
Renal Clearance (CLr) of Metformin in the Presence and Absence of VX-993 | From Day 1 up to Day 14
Metformin Fraction Excreted Unchanged (fe) in Urine in the Presence and Absence of VX-993 | From Day 1 up to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing